CLINICAL TRIAL: NCT06908681
Title: Impact of Intertransverse Process Block on Postoperative Acute Pain in Patients Undergoing Coronary Artery Bypass Grafting Via Median Sternotomy: A Prospective, Randomized Controlled Trial"
Brief Title: Intertransverse Process Block for Postoperative Acute Pain After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Aydemir (Other)
Collaborators: Konya City Hospital (Other)
Responsible Party: Sponsor-Investigator, Mustafa Aydemir, Specialist, Department of Anesthesiology and Reanimation, Konya City Hospital
Organization: Konya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSTF-KVCAGRI-2025-01
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Coronary Artery Bypass Grafting (CABG) Surgery; Sternotomy
Keywords: Intertransverse Process Block; Coronary Artery Bypass Grafting; Postoperative Pain; Cardiac Surgery; Median Sternotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group receiving bilateral intertransverse process block (ITPB) with 0.25% bupivacaine, or the control group receiving saline injection at the same anatomical site. Each participant will receive only one type of intervention. The study is designed as a parallel, triple-blind, randomized controlled trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study uses a triple-blind design. Participants, the anesthesiologist performing the block, and the investigators assessing postoperative outcomes are blinded to group allocation. The person preparing the injection syringes is not involved in patient care or outcome assessment, ensuring proper concealment of group assignments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITPB Group (Experimental): Patients in this group will receive a bilateral intertransverse process block (ITPB) with 0.25% bupivacaine (20 mL per side) under ultrasound guidance before coronary artery bypass grafting.
  Interventions: Procedure: Bilateral Intertransverse Process Block (ITPB)
- Control Group (Placebo Comparator): Patients in this group will receive bilateral saline injections (20 mL per side) at the same anatomical site under ultrasound guidance prior to surgery.
  Interventions: Procedure: placebo saline injection

INTERVENTIONS:
Procedure: Bilateral Intertransverse Process Block (ITPB) — A bilateral intertransverse process block (ITPB) will be performed under ultrasound guidance using 20 mL of 0.25% bupivacaine per side prior to coronary artery bypass grafting. The block targets the dorsal rami of thoracic spinal nerves to provide postoperative analgesia.
  Arms: ITPB Group
Procedure: placebo saline injection — A bilateral placebo injection (20 mL of 0.9% saline per side) will be administered at the same anatomical site under ultrasound guidance prior to coronary artery bypass grafting, mimicking the ITPB procedure without active drug.
  Arms: Control Group

SUMMARY:
This prospective, randomized controlled trial aims to evaluate the effect of bilateral intertransverse process block (ITPB) on acute postoperative pain in patients undergoing coronary artery bypass grafting (CABG) via median sternotomy. Patients will be randomly assigned to receive either ITPB or placebo (saline) injection prior to surgery. Postoperative pain scores, opioid consumption, and recovery quality will be assessed during the first 24 hours following extubation.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is associated with significant postoperative pain due to sternotomy and tissue manipulation, which may impair recovery, increase opioid consumption, and prolong hospital stay. Regional anesthesia techniques are increasingly used as part of multimodal analgesia strategies to minimize opioid-related side effects. The intertransverse process block (ITPB) is a novel regional technique that targets the dorsal rami of spinal nerves and may provide effective bilateral analgesia in thoracic procedures with a favorable safety profile.

This prospective, randomized, triple-blind controlled study aims to investigate the effect of preoperative bilateral ITPB on postoperative acute pain, opioid consumption, and recovery quality in adult patients undergoing elective CABG via median sternotomy. Patients will be randomized to receive either ITPB with 0.25% bupivacaine or a placebo (saline) injection under ultrasound guidance. Postoperative outcomes, including Numeric Rating Scale (NRS) pain scores, rescue analgesic use, total opioid consumption, and Quality of Recovery-15 (QoR-15) scores, will be collected within the first 24 hours following extubation. The results of this study may support the incorporation of ITPB into routine analgesia protocols for cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective coronary artery bypass grafting (CABG) via median sternotomy planned
* Able to provide written informed consent
* Able to communicate symptoms reliably with the research team

Exclusion Criteria:

* Emergency CABG surgery
* Infection or open wound at the injection site
* Coagulopathy
* Hepatic or renal failure
* Reoperation cases
* Incomplete or missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores at 0, 6, 12, and 24 Hours After Extubation | Within 24 hours after extubation
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), a numerical scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain. Scores will be recorded at 0, 6, 12, and 24 hours following extubation.

SECONDARY OUTCOMES:
Total Opioid Consumption in the First 24 Hours Postoperatively | Within 24 hours after extubation
  The total amount of opioids administered will be calculated in milligrams of morphine equivalents (mg MEQ) from extubation until the 24th postoperative hour.
Number of Patients Requiring Rescue Analgesia | Within 24 hours after extubation
  The number of patients who require intravenous tramadol 100 mg due to a Numeric Rating Scale (NRS) score greater than 4 within the first 24 hours will be recorded.
Quality of Recovery Score (QoR-15) at 24 Hours Postoperatively | 24 hours after extubation
  The Turkish version of the Quality of Recovery-15 (QoR-15) questionnaire will be administered 24 hours after extubation to assess overall postoperative recovery. The scale ranges from 0 to 150, and higher scores indicate better recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to institutional policies and ethical considerations regarding patient confidentiality.